CLINICAL TRIAL: NCT03795480
Title: A Randomized-controlled Trial (RCT) on the Efficacy of a New Online Intervention for Depression: MOOD
Brief Title: Online Intervention for Depression: MOOD
Acronym: MOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOOD
Record Dates: First submitted 2018-08-16; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOOD (Experimental): The online program "MOOD" is based on methods of cognitive behavior therapy (KVT) and contains elements of mindfulness and metacognition. Participants can contact a moderator (trained psychologists) if they have any questions. However, this function is optional. The program consists of nine interactive modules, one of which is an introductory module. The other modules are called: ABC-Scheme, Positive Activities, Self-Worth, Social Competence, Mindfulness, Modifying Thoughts, Sleep, and Relapse Prevention.
  Interventions: Behavioral: MOOD
- Control (No Intervention): The wait-list control group does not receive additional treatment. However, previously started therapies (psychotherapy/ psychopharmacotherapy) may be continued during the study. Individuals of the wait-list control group receive access to MOOD after completion of the post-assessment.

INTERVENTIONS:
Behavioral: MOOD — MOOD is an online self-help program targeted on depressive symptoms. The program consists of nine modules, one of which is an introductory module. The other modules are called: ABC-Scheme, Positive Activities, Self-Worth, Social Competence, Mindfulness, Modifying Thoughts, Sleep, and Relapse Prevention. All modules are based on principles of cognitive behavioral therapy (CBT) and include elements of mindfulness-based and metacognitive techniques. The modules contain interactive exercises which are aimed at incorporating the participant's experiences into the program and increasing identification of the participant with the presented material. Participants are free to work through the different modules in their own speed and way, however, it is recommended to work on one to two modules per week.
  Arms: MOOD

SUMMARY:
The study aims to examine the efficacy and acceptance of a self-help internet intervention "MOOD" in a sample of individuals with depressive symptoms. It is tested whether depressive symptomatology decreases in the intervention group compared to a wait-list control group. Further aims are to ascertain changes in self-worth and quality of life, to assess subjective evaluation of the program and to examine whether expectations of the program's helpfulness would predict symptom reduction.

DETAILED DESCRIPTION:
The study aims to examine the efficacy and acceptance of a self-help internet intervention "MOOD" in a sample of individuals with depressive symptoms. It is tested whether depressive symptomatology decreases in the intervention group compared to a wait-list control group. Secondary aims are to ascertain changes in self-worth and quality of life, to assess subjective evaluation of the program and to examine whether expectations of the program's helpfulness would predict symptom reduction. During the intervention period of six weeks, participants of the intervention group have access to the online program MOOD. Prior and following this period both groups complete a pre- and post-assessment. Participants of the wait-list control group receive access to MOOD following the post-assessment.

ELIGIBILITY:
Inclusion Criteria:

* presence of psychological strain and desire for treatment for depressive symptoms
* internet access
* sufficient command of the German language

Exclusion Criteria:

* acute suicidality (as assessed with one item of the BDI)
* lifetime diagnoses of bipolar disorder and psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2018-07-22 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | Change in BDI from baseline to post (intervention period is 6 weeks)
  This questionnaire assesses symptoms of depression and their severity (Beck, Steer, & Brown, 1996). It contains 21 items and the participant is asked to rate how severe he or she experiences each symptom on a 4-point Likert scale ranging from 0 (not at all severe) to 3 (extreme form of each symptom).

SECONDARY OUTCOMES:
Rosenberg self-esteem scale (RSE) | Change in RSE from baseline to post (intervention period is 6 weeks)
  The RSE is a self-report questionnaire assessing an individual's self-esteem (Rosenberg, 1965) The scale consists of 10 items and the participants are asked to rate in how far they agree with each item on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree".
WHOQOL-Bref | Change in WHOQOL-Bref from baseline to post (intervention period is 6 weeks)
  The WHOQOL-Bref is a questionnaire assessing Quality of Life (QOL) (Whoqol Group, 1998). It is an abbreviated version of the WHOQOL-100 and contains 26 items. The questionnaire has four types of 5-point Likert scales asking the participant "how much", "how completely", "how often", "how good" or "how satisfied" he felt in the last two weeks. The four different scales are distributed across the four domains sampled in this questionnaire: Physical health, Psychological, Social relations, Environment.
University of Rhode Island Change Assessment (URICA) | Only at Baseline (pre intervention)
  The URICA is a measure of willingness to change (Dozois, Westra, Collins, Fung & Garry, 2004) and was assessed at baseline. It consists of 32 items that depict four stages of change: pre-contemplation, contemplation, action and maintenance. In the present study, in total 9 items are used which were chosen from the subscales of pre-contemplation, contemplation and action. Internal consistency is .83 and test-retest reliability lies between .63-.75.
Subjective appraisal | Only at post-assessment (6 weeks)
  In the post-assessment, individuals of the intervention group also answered questions on subjective evaluation and appraisal of the program. Items were for example "I think this program is useful as a self-help tool" or "I had to bring myself to make use of the program". The items could be answered on a 4-point Likert scale ranging from "Totally disagree" to "Totally agree". Participants also had the possibility to provide feedback on the program.
Patient Health Questionnaire-9 Depression Module (PHQ-9) | Change in PHQ-9 from baseline to post (intervention period is 6 weeks)
  The PHQ-9 is used to measure depression and its severity (Kroenke, Spitzer, & Williams, 2001). It consists of 9 items which can be rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day), depending on the severity and frequency of the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Moritz, Prof., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department for Psychiatry and Psychotherapy of University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bucker L, Schnakenberg P, Karyotaki E, Moritz S, Westermann S. Diminishing Effects After Recurrent Use of Self-Guided Internet-Based Interventions in Depression: Randomized Controlled Trial. J Med Internet Res. 2019 Oct 2;21(10):e14240. doi: 10.2196/14240. PMID 31579014